CLINICAL TRIAL: NCT07101588
Title: Ruxolitinib and Decitabine-Enhanced Conditioning Versus Modified Bu/Cy or BuF Conditioning for the Impact on Relapse of Acute Myeloid Leukemia in First Complete Remission (CR1)After Allogeneic Hematopoietic Stem Cell Transplantation: A Multicenter, Prospective Randomized Controlled Trial
Brief Title: Ruxolitinib-Decitabine Intensified Conditioning Regimen for AML: A Randomized Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University, Zhengzhou (Unknown); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Dr., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2024-678-01
Record Dates: First submitted 2025-06-01; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: HSCT
MeSH Terms: interventions — ruxolitinib; Decitabine

STUDY DESIGN:
Intervention Model Description: Random Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Interventions (Active Comparator): 1. Decitabine: 20 mg/m²/day, administered from Day -15 to Day -10.
  2. Ruxolitinib(with Voriconazole):
     * 10 mg twice daily (bid), Day -15 to Day -5
     * 5 mg twice daily (bid), Day -4 to Day -3
     * 5 mg once daily (Qd), Day -2
  3. Busulfan (Bu): 0.8 mg/kg every 6 hours (Q6h), Day -8 to Day -6.
  4. Carmustine (BCNU): 250 mg every 8 hours (Q8h), Day -3.
  5. Cytarabine (Ara-C):
     * 4 g/m²/day, Day -10 to Day -9 (for unrelated or haploidentical donors)
     * 4 g/m²/day, Day -9 only (for matched sibling donors)
  6. Cyclophosphamide (CTX): 50 mg/kg/day, Day -5 to Day -4. or Fludarabine 30mg/m2/day, iv, Day -6 to Day -2;
  7. Antithymocyte Globulin (ATG):
     * 10 mg/kg/day, Day -5 to Day -2 (for unrelated or haploidentical donors)
     * 5 mg/kg/day, Day -5 to Day -2 (for matched sibling donors)
  Interventions: Combination Product: Ruxolitinib, Decitabine
- The control group (No Intervention): 1. Busulfan (Bu): 0.8 mg/kg every 6 hours (Q6h), Day -8 to Day -6.
  2. Carmustine (BCNU): 250 mg every 8 hours (Q8h), Day -3.
  3. Cytarabine (Ara-C):
     * 4 g/m²/day, Day -10 to Day -9 (for unrelated or haploidentical donors)
     * 4 g/m²/day, Day -9 only (for matched sibling donors)
  4. Cyclophosphamide (CTX): 50 mg/kg/day, Day -5 to Day -4. or Fludarabine 30mg/m2/day, iv, Day -6 to Day -2;
  5. Antithymocyte Globulin (ATG):
     * 10 mg/kg/day, Day -5 to Day -2 (for unrelated or haploidentical donors)
     * 5 mg/kg/day, Day -5 to Day -2 (for matched sibling donors)

INTERVENTIONS:
Combination Product: Ruxolitinib, Decitabine — 1. Decitabine: 20 mg/m²/day, administered from Day -15 to Day -10.
  2. Ruxolitinib:
     * 10 mg twice daily (bid), Day -15 to Day -5
     * 5 mg twice daily (bid), Day -4 to Day -3
     * 5 mg once daily (Qd), Day -2
  Arms: Assigned Interventions

SUMMARY:
This study aims to determine whether the recurrence rate of high-risk acute myeloid leukemia CR1 patients who received allogeneic hematopoietic stem cell transplantation with the Ruxolitinib, Decitabine combined with Bu/Cy or BuF intensive pretreatment regimen is reduced compared with the traditional Bu/Cy or BuFpretreatment regimen.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation is the only radical treatment for high-risk acute myeloid leukemia (AML), but the traditional Bu/Cy pretreatment regimen is highly toxic and has a high recurrence rate after transplantation (the long-term survival rate is only 10-30%). Although the existing improved regimens such as sequential chemotherapy can reduce the leukemia burden, they lead to prolonged myelosuppression time (17-39 days) and a non-relapse mortality rate as high as 17.2%. There is an urgent need to develop new pretreatment regimens that have both strong anti-leukemia effects and low toxicity.

Studies have found that the JAK-STAT signaling pathway is generally abnormally activated in hematological tumors such as AML. The objective response rate of Ruxolitinib (a JAK1/2 inhibitor) as a monotherapy for relapsed/refractory leukemia reached 45%. When combined with the demethylated drug decitabine, it can synergistically inhibit leukemia cells. Clinical data show that decitabine reduces the recurrence rate after transplantation by 20% (15.0% vs 38.3%), and the combination of the two has good safety. The main adverse reaction is grade 1-2 hematological toxicity.

Our center innovatively proposed the Rux-Dec-mBu/Cy or BuF combined regimen: integrating Ruxolitinib (step-based dose reduction) and decitabine (20mg/m²/d) on the basis of the classic Bu/Cy or BuF. Previous single-arm studies have shown that the one-year recurrence rate of CR1 patients is 0%, and the incidence of toxicity above grade 3 is less than 11%. This study intends to conduct a multicenter randomized controlled trial to verify the superiority of this regimen in reducing recurrence after transplantation in patients with high-risk AML CR1. Its core advantage lies in simultaneously achieving anti-leukemia enhancement (through JAK-STAT targeting and epigenetic regulation) and controllable toxicity (The median grain deficiency time was shortened to 14 days).

ELIGIBILITY:
Inclusion Criteria:

* 1) Acute myeloid leukemia with indications for allogeneic hematopoietic stem cell transplantation, CR1 2) Have HLA-matched sibling donors or haploidentical donors or ≥8/10 HLA-matched unrelated donors 3) The patients' ages range from 12 to 64 years old 4) Liver function: ALT and AST≤2.5 times the upper limit of normal values, bilirubin ≤2 times the upper limit of normal values 5) Renal function: Creatinine ≤ the upper limit of the normal value 6) There are no uncontrollable infections or serious mental and psychological disorders 7) Sign the informed consent form.

Exclusion Criteria:

* 1. Patients with acute promyelocytic leukemia (M3) 2. One of the donor and recipient is pregnant 3. Suffering from mental illness or other conditions that prevent one from following the plan.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
GRFS | 1 year
  GVHD-free, relapse-free survival (GRFS) was defined as a composite endpoint of death from any cause, disease relapse, grade Ⅲ-Ⅳ acute GVHD, or chronic GVHD requiring systemic immunosuppression therapy.

SECONDARY OUTCOMES:
Cumulative recurrence rate (CIR) | 1 years after transplantation
  Calculated from the first day after stem cell infusion to the last follow-up, the number of patients with hematological or MRD recurrence/the total number of cases ×100%. The definition of hematological recurrence: After remission, patients present with one of the following three conditions: (1) ≥5% of primary lymphocytes and immature lymphocytes in the bone marrow; (2) Extramedullary leukemia occurs; (3) Leukemia cells were found in peripheral blood smears. The definition of MRD recurrence: Leukemia cells are detected by flow cytometry or molecular biology.
Progression-Free Survival（PFS） | 1 years after transplantation
  The time from the date of transplantation to the recurrence of leukemia or death for any reason.
CR rate | 30 days after transplantation
  The proportion of bone marrow in complete remission from the first day after stem cell infusion to +30 days.
The incidence of aGVHD | 100 days after transplantation
  Calculated from the first day after stem cell infusion, the time from the occurrence of aGVHD, the time of recurrence or death. The actual incidence rate is the number of patients who occur/the total number of cases ×100%.
The incidence of cGVHD | 1 years after transplantation
  Calculated from the first day after stem cell infusion, the time from the occurrence of cGVHD, the time of recurrence or death. The actual incidence rate is the number of patients who occur/the total number of cases ×100%.
Disease-free survival rate (DFS) | 1 years after transplantation
  Disease-free survival rate (DFS) refers to the survival period without evidence of recurrence or progression.
Treatment-related safety indicators | 1 years after transplantation
  Mainly include bacterial infection, viral infection, fungal infection, and PTLD from the time calculated after transplantation to the last follow-up.
Non-relapse mortality | 1 year
  Non-relapse mortality (NRM) was defined as death from any cause other than disease relapse.
The cumulative incidence of virus reactivation | Day +180 days post-transplantation
  The cumulative incidence of virus reactivation by Day +180 days post-transplantation was defined as the proportion of virus reactivation occurring at any monitoring point during days 180 post-transplant.
Graft failure | +28 days after transplantation
  Graft failure was defined as non-engraftment (ie, autologous reconstitution) or graft rejection (ie, secondary loss of donor chimerism) at +28 days
Neutrophil engraftment | +28 days after transplantation
  Neutrophil engraftment was defined as the first of three consecutive days with a neutrophil count >0.5 ×109/L.
Platelet engraftment | +28 days after transplantation
  Platelet engraftment was defined as the first of seven consecutive days with a platelet count >20×109/L without transfusion support.
CD4+T cell reconstitution | the first 100 days post-transplantation
  CD4+T cell reconstitution was defined as CD4+ T cell count ≥ 50/μL in two consecutive measurements within the first 100 days post-transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data contain sensitive personal health information

REFERENCES:
- [Background] Xuan L, Dai M, Jiang E, Wang Y, Huang F, Fan Z, Xu N, Nie D, Liang X, Chen H, Ye J, Shi P, Liu H, Jin H, Lin R, Yan C, Zhang Y, Sun J, Han M, Liu Q. The effect of granulocyte-colony stimulating factor, decitabine, and busulfan-cyclophosphamide versus busulfan-cyclophosphamide conditioning on relapse in patients with myelodysplastic syndrome or secondary acute myeloid leukaemia evolving from myelodysplastic syndrome undergoing allogeneic haematopoietic stem-cell transplantation: an open-label, multicentre, randomised, phase 3 trial. Lancet Haematol. 2023 Mar;10(3):e178-e190. doi: 10.1016/S2352-3026(22)00375-1. Epub 2023 Jan 23. PMID 36702138
- [Background] Li Z, Shi W, Lu X, Lu H, Cao X, Tang L, Yan H, Zhong Z, You Y, Xia L, Hu Y, Wang H. Decitabine-Intensified Modified Busulfan/Cyclophosphamide Conditioning Regimen Improves Survival in Acute Myeloid Leukemia Patients Undergoing Related Donor Hematopoietic Stem Cell Transplantation: A Propensity Score Matched Analysis. Front Oncol. 2022 Mar 16;12:844937. doi: 10.3389/fonc.2022.844937. eCollection 2022. PMID 35371981
- [Background] Watanabe T. [Drug tolerance in microorganisms, with special reference to genetic study of its transmission]. Nihon Saikingaku Zasshi. 1969 Oct;24(9):418-25. No abstract available. Japanese. PMID 4908810
- [Background] Tang X, Valdez BC, Ma Y, Zhang Q, Qu C, Dai H, Yin J, Li Z, Xu T, Xu Y, Chen J, Zhu X, Chen Z, Wu D, Andersson BS. Low-dose decitabine as part of a modified Bu-Cy conditioning regimen improves survival in AML patients with active disease undergoing allogeneic hematopoietic stem cell transplantation. Bone Marrow Transplant. 2021 Jul;56(7):1674-1682. doi: 10.1038/s41409-021-01238-5. Epub 2021 Feb 26. PMID 33637882
- [Background] Tsukada T, Fukushima M, Takebe H, Nakai Y. Vasoactive intestinal peptide gene expression in the rat pheochromocytoma cell line PC12. Mol Cell Endocrinol. 1995 Feb;107(2):231-9. doi: 10.1016/0303-7207(94)03448-3. PMID 7768335
- [Background] Schmid C, Schleuning M, Schwerdtfeger R, Hertenstein B, Mischak-Weissinger E, Bunjes D, Harsdorf SV, Scheid C, Holtick U, Greinix H, Keil F, Schneider B, Sandherr M, Bug G, Tischer J, Ledderose G, Hallek M, Hiddemann W, Kolb HJ. Long-term survival in refractory acute myeloid leukemia after sequential treatment with chemotherapy and reduced-intensity conditioning for allogeneic stem cell transplantation. Blood. 2006 Aug 1;108(3):1092-9. doi: 10.1182/blood-2005-10-4165. Epub 2006 Mar 21. PMID 16551971
- [Background] Pankhurst R. The earliest history of famine and pestilence in Ethiopia and a note on the "Egyptian Deaths" of 17th and 18th century Ethiopia. Ethiop Med J. 1973 Jul;11(3):233-6. No abstract available. PMID 4602511
- [Background] Thomas HC, McSween RN, White RG. Role of the liver in controlling the immunogenicity of commensal bacteria in the gut. Lancet. 1973 Jun 9;1(7815):1288-91. doi: 10.1016/s0140-6736(73)91300-7. No abstract available. PMID 4126078
- [Background] Camera A, Rinaldi CR, Palmieri S, Cantore N, Mele G, Mettivier V, Miraglia E, Mastrullo L, Grimaldi F, Luciano L, Guerriero A, Rotoli B, Ferrara F. Sequential continuous infusion of fludarabine and cytarabine associated with liposomal daunorubicin (DaunoXome) (FLAD) in primary refractory or relapsed adult acute myeloid leukemia patients. Ann Hematol. 2009 Feb;88(2):151-8. doi: 10.1007/s00277-008-0571-z. Epub 2008 Aug 16. PMID 18709502
- [Background] Fiegl M, Unterhalt M, Kern W, Braess J, Spiekermann K, Staib P, Gruneisen A, Wormann B, Schondube D, Serve H, Reichle A, Hentrich M, Schiel X, Sauerland C, Heinecke A, Rieger C, Beelen D, Berdel WE, Buchner T, Hiddemann W; German AML Cooperative Group (AMLCG). Chemomodulation of sequential high-dose cytarabine by fludarabine in relapsed or refractory acute myeloid leukemia: a randomized trial of the AMLCG. Leukemia. 2014 May;28(5):1001-7. doi: 10.1038/leu.2013.297. Epub 2013 Oct 22. PMID 24150216